**Tazarotene Cream 0.1%** 

Protocol /

0454-01-01/

# STATISTICAL ANALYSIS PLAN

A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.1% to TAZORAC® (Tazarotene) Cream 0.1% and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris

Protocol Number: 0454-01-01 / NCT02886715

# **Sponsor:**

Fougera Pharmaceuticals Inc. 60 Baylis Road Melville, New York, 11747

**Contract Research Organization:** 

April 26, 2017

Final Version 2.0

**Tazarotene Cream 0.1%** 

Protocol /

0454-01-01/

# SAP FINAL VERSION APPROVALS

A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.1% to TAZORAC® (Tazarotene) Cream 0.1% and Both Active Treatments to a Vehicle Control in the Treatment of Acne Vulgaris

| Written By: | |
|--------------|-------|
| Signature: | Date: |
| Reviewed By: | |
| Signature: | Date: |
| Approved By: | |
| Signature: | Date: |

Tazarotene Cream 0.1% Protocol / 0454-01-01/

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---------|------|--------------------------|------------|

Tazarotene Cream 0.1%

Protocol /

0454-01-01/

## List of Abbreviations and Definition of Terms

ADaM Analysis Data Model

AE Adverse Event

ANOVA Analysis of Variance

C Celsius

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval CRF Case Report Form

CRO Contract Research Organization eCRF Electronic Case Report Form

EOS End of Study Fahrenheit

FDA Food and Drug Administration GLM Generalized Linear Model

Hg Mercury

ICF Informed Consent Form

ICH International Conference on Harmonisation

IGA Investigator Global Assessment

IP Investigational Product

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

mITT modified Intent-to-Treat Population

OGD Office of Generic Drugs PD Protocol Deviation

PP Per-Protocol PROC Procedure

RLD Reference Listed Drug
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System

SD Standard Deviation

SDTM Study Data Tabulation Model

# **TABLE OF CONTENTS**

| 1. INTRODUCTION | |
|---|---|
| 2. OBJECTIVES | |
| 3. OVERALL STUDY DESIGN | |
| 4. RANDOMIZATION AND BLINDING | 11 |
| 5. SAMPLE SIZE | |
| 6. ANALYSIS POPULATION | |
| 7. STUDY EFFICACY VARIABLES | 13 |
| 8. STATISTICAL ANALYSIS METHODS | 14 |
| 8.1 Baseline Characteristics | 14 |
| 8.1.1 Demographics Comparability of Treatment Groups | 14 |
| 8.1.2 Medical History | |
| 8.1.3 Concomitant Medications | 15 |
| 8.1.4 Pregnancy Test | 15 |
| 8.2 Efficacy Analyses | 15 |
| 8.2.1 Primary Efficacy Analysis | |
| 8.2.2 Secondary Efficacy Analyses | |
| 8.2.3 Treatment-by-Site Interaction and Pooling of Clinical Sites | |
| 8.3 Safety Analysis | |
| 8.3.1 Adverse Events | |
| 8.3.2 Application Site Reactions | |
| 8.3.3 Vital Signs | |
| 8.4 Multiple Comparisons | |
| 8.5 Methods for Handling Missing Data | |
| 8.6 Interim Analyses | |
| 9. TABLE, LISTING AND FIGURE SHELLS | |
| T16.1.9.1 Summary of Discontinued Subjects (Safety Population) | |
| T16.1.9.2 Summary of Protocol Deviations (Safety Population) | |
| T16.1.9.3.1 Summary of Subjects Excluded from Efficacy Analysis | |
| T16.1.9.3.2 Summary of Subjects Included in Analysis Population by Study Cer | |
| T16.1.9.4.1 Summary of Demographic Data (Safety Population) | 26 |
| T16.1.9.5.1 Summary of Demographic Data (modified Intent-to-Treat Populat | ion). 28 |
| T16.1.9.5.2 Summary of Baseline Parameters (modified Intent-to-Treat Popula | |
| T16.1.9.6.1 Summary of Demographic Data (Per-Protocol Population) | 28 |
| T16.1.9.6.2 Summary of Baseline Parameters (Per-Protocol Population) | |
| T16.1.9.7.1 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent C | |
| Baseline in Inflammatory Lesion Count) (Per-Protocol Population) | |
| T16.1.9.7.2 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent C | |
| | 0 |
| Baseline in Inflammatory Lesion Count) (modified Intent-to-Treat Pop | |
| T16.1.9.8.1 Summary of Analysis Results of Co-Primary Efficacy Endpoint | 31 |
| T16.1.9.8.2 Summary of Supportive Analysis Results of Co-Primary Efficacy E | ndpoint |
| 2 control of the property of t | 32 |
| T16.1.9.9.1 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent C | |
| Baseline in Non-Inflammatory Lesion Count) (Per-Protocol Population | 1) 33 |

| Tazarotene Cream 0.1% | Protocol / | 0454-01-01/ |
|---|---|---|
| T16.1.9.9.2 Descriptive Summary of Co-F<br>Baseline in Non-Inflammatory Lo | | |
| Population) | * * | |
| T16.1.9.10.1 Summary of Analysis Result | | |
| T16.1.9.10.2 Summary of Supportive Ana | | |
| <b>T16.1.9.11 Summary of Analysis Results</b> | of Secondary Efficacy En | dpoint 37 |
| T16.1.9.12 Overall Summary of Adverse | | |
| T16.1.9.13 Summary of Frequency of All Population) | <b>Adverse Events by Body</b> | System (Safety |
| T16.1.9.14 Summary of Frequency for Al System (Safety Population) | | |
| T16.1.9.15 Summary of Frequency of All | <b>Adverse Events by Severi</b> | ity (Safety Population) |
| T16.1.9.16 Summary of Frequency of All Population) | <b>Adverse Events by Relati</b> | onship (Safety |
| T16.1.9.17 Summary of Frequency of Ser | | |
| T16.1.9.18 Summary of Application Site | | |
| T16.1.9.19 Summary of Frequency of Ap | | |
| T16.1.9.20 Summary of Vital Signs (Safe | | |
| L16.2.1 Listing of Discontinued Subjects. | | |
| L16.2.2 Listing of Protocol Deviations | | |
| L16.2.3.1 Subjects Excluded from the Per | | |
| L16.2.3.2 Subjects Excluded from the Mo | | |
| L16.2.4.1 Listing of Demographic Data | | |
| L16.2.4.2 Listing of Medical History | | |
| L16.2.4.3 Listing of Concomitant Medica | | |
| L16.2.5.1 Listing of Visit Date Information | | |
| L16.2.5.2 Listing of Drug Administration | | |
| L16.2.6.1 Listing of Lesion Count | | |
| L16.2.6.2 Listing of Investigator Global A | | |
| L16.2.7.1 Listing of Adverse Events by The | | |
| L16.2.7.2 Listing of Application Site Read | | |
| L16.2.8.1 Listing of Pregnancy Test Resu | lts | 59 |
| L16.2.8.2 Listing of Vital Signs | | |
| APPENDIX A: Investigator's Global Asses | | |
| APPENDIX B: Application Site Reactions. | | |

63

**Tazarotene Cream 0.1%** 

Protocol /

0454-01-01/

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 0454-01-01 Rev. 2 dated 12/22/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol 0454-01-01 Rev. 2 dated 12/22/2016
- Final eCRF Version 1.0 for

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

## 2. OBJECTIVES

The objectives of this study are to:

- 1. Evaluate the therapeutic equivalence of the Test product, Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) to the Reference product, TAZORAC® (tazarotene) Cream 0.1% (Allergan, Inc.) in the treatment of acne vulgaris.
- 2. Demonstrate the superiority of the efficacy of the Test and Reference (active) products over that of the Placebo in the treatment of acne vulgaris.
- 3. Compare the safety of the Test, Reference and Placebo products in the treatment of acne vulgaris.

#### 3. OVERALL STUDY DESIGN

This multi-center, double-blind, randomized, vehicle-controlled, parallel-group bioequivalence clinical study has been designed to evaluate the efficacy and safety of a generic tazarotene cream

## **Tazarotene Cream 0.1%**

Protocol /

0454-01-01/

0.1% (Fougera Pharmaceuticals Inc.) compared to the FDA Reference Listed Drug (RLD) TAZORAC® (tazarotene) Cream, 0.1% (Allergan) in subjects with a clinical diagnosis of acne vulgaris. Additionally, both the Test product and Reference (i.e., the RLD) product will be tested for superiority to a Placebo. Subjects with confirmed facial acne vulgaris will apply the investigational product (IP) once daily, in the evening, for 84 days  $\pm$  4 days (12 weeks).

Before any study-specific procedures are performed, all subjects will read and sign the IRB-approved ICF. For a subject considered to be a minor in the state he/she is screened, the parent or legal guardian will be required to sign the ICF and the subject will sign an IRB-approved "assent to participate" form, as applicable.

Each site will develop an individualized recruitment plan to collectively enroll approximately 1110 eligible subjects,  $\geq 12$  to  $\leq 40$  years of age, with a clinical diagnosis of acne vulgaris and meeting the inclusion/exclusion criteria. Subjects will be randomized to one of the three IPs as follows:

- Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)
- Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)
- Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Subjects will attend the following scheduled clinic visits:

- Visit 1 Screening/Baseline: Day -14 to 1
- Visit 2 Interim Visit: Day  $28 \pm 4$  days
- Visit 3 Interim Visit: Day  $56 \pm 4$  days
- Visit 4 End of Study: Day  $85 \pm 4$  days

Subjects may attend unscheduled clinic visits:

• Visit 9999 – Unscheduled visit

At Visit 1, eligible subjects will be randomized to the Test, Reference or Placebo product in a 2:2:1 ratio using which is an interactive response technology (IRT) system provided by the IRT provider. Study subjects will be provided with of IP. At Visit 2 and/or Visit 3, subjects who continue to be eligible for continuation in the study can be dispensed another of investigational product, as needed, based on the amount of IP remaining from the tube previously dispensed. Further, any empty tubes will be collect at these visits. At Visit 4, all tubes will be collected (used and unused). A subject may return for an Unscheduled Visit at any time, should they require a resupply of IP (i.e., tube lost; all IP used between visits). It is estimated that up to will be needed to dose the subject for the treatment period. Additional tubes beyond the initial will only be dispensed if the initial supply is lost and/or significantly damaged (i.e., becomes punctured) and warrants replacement.

Tazarotene Cream 0.1% Protocol / 0454-01-01/

The day that the subject administers their first dose of IP will be considered Day 1.

For all other subjects, the first

dose (Day 1) of IP will be applied on the evening of Visit 1.

The subject will be instructed to apply a thin layer  $(2 \text{ mg/cm}^2)$  of the product once daily, in the evening, through the evening before Visit 4 (Day  $85 \pm 4$ ). There will be no application of the product on the day of the End of Study visit.

Efficacy evaluations will be based on dermatological assessments in the clinic. The two co-primary statistical analyses of interest are (1) the percent change from Baseline to Week 12 in the inflammatory (papules/pustules) lesion counts and (2) the percent change from Baseline to Week 12 in the non-inflammatory (open and closed comedones) lesion counts. The secondary analysis is the proportion of subjects who are considered a Clinical Success at Week 12, as defined by an IGA score that is at least 2 grades less than the Baseline assessment. A Clinical Failure is defined as an IGA score that is the same, higher or one grade lower than the Baseline IGA at Week 12 (Appendix A).

**Tazarotene Cream 0.1%** 

Protocol /

0454-01-01/

# **Study Schematic**

| PROCEDURE | VISIT 1<br>(Day -14 to 1)<br>Screening/<br>Baseline | VISIT 2<br>(Day 28<br>± 4 Days)<br>Interim Visit | VISIT 3<br>(Day 56<br>± 4 Days)<br>Interim Visit | VISIT 4 (Day 85 ± 4 Days)* End of Study/ Early Termination |
|---|---|---|---|---|
| Informed Consent/Assent | X <sup>‡</sup> | | | |
| Medical History/<br>Demographics | X <sup>‡</sup> | | | |
| Pregnancy Test <sup>†</sup> | X <sup>‡</sup> | X | X | X |
| Vital Signs | $X^{\ddagger}$ | | | X |
| Lesion Counts | X <sup>‡</sup> | X | X | X |
| Investigator's Global<br>Assessment | X <sup>‡</sup> | X | X | X |
| Application Site Reactions | X | X | X | X |
| Inclusion/Exclusion<br>Criteria Review | X <sup>‡</sup> | | | |
| Concomitant Medication | X <sup>‡</sup> | X | X | X |
| Randomization | X | | | |
| Dispense IP | X | X** | X** | |
| Return of IP | | X** | X** | X |
| Dispense Subject Diary /Supplies | X | X | X | |
| Collect/Review Subject<br>Diary | | X | X | X |
| Adverse Events | | X | X | X |
| Discharge from Study | | | | X |

<sup>\*</sup> Dosing regimen is once daily in the evening through the evening for 84 days (Day 1 to Day 84) before Visit 4 (Day  $85 \pm 4$ )

<sup>\*\*</sup> If applicable, based on use of previously dispensed product.

<sup>†</sup> For females of childbearing potential

<sup>‡</sup> Procedures performed as part of the screening assessment, before randomization

Tazarotene Cream 0.1% 0454-01-01/ Protocol / 4. RANDOMIZATION AND BLINDING The IP will be randomized, packaged and blinded by an . The randomization code will be generated using a validated computer program. Each site will receive multiple, full blocks of IP in each delivery. The quantity received may vary. Randomization will be pre-planned according to a computer-generated randomization scheme. The randomization code will be retained within which is maintained by will also retain the kit boxes numbers supplied to each site and the kit boxes numbers that have been selected for retention and are therefore unavailable for dispensing to subjects. Upon confirmation of subject eligibility, the subject's information (i.e., subject's initials, date of , and the system will assign a birth, etc.) will be entered into randomization number to the subject based upon will then assign the subject a kit box number in a blinded fashion at Visit 1. This kit box number will correspond to a specific treatment group within some specific treatment group will be unknown to the Investigator, the CRO, the sponsor and the subject. The site will record the randomization number and the kit box number in the subject's source documentation and drug will then dispense dispensing log. The from the kit box. The will record the tube number of the dispensed to the subject in the subject's source documentation and drug dispensing log. At Visits 2, 3 and/or Unscheduled Visit, additional IP may be dispensed to the subject, as needed. The an additional unused tube from the subject's previously assigned kit box, dispense it to the subject and record the tube number. Each subject will maintain the same treatment assignment throughout the study. **5. SAMPLE SIZE** Sample size calculations were performed using For the primary endpoint analysis (percent change from Baseline at Week 12 (Study Day 85 ± 4 days) in

sample size estimations are based on data reported in the

inflammatory and non- inflammatory lesion counts), the sample size is estimated for therapeutic equivalence of the Test to the Reference product and superiority of each of the active treatments groups over Placebo. As no variability data were available for TAZORAC® Cream, 0.1%, the

| ester to be approximately exercised to be approximately exercised approximately exercised approximately exercised equivalence limits. | flammatory lesion count attely with a SD of subjects per power to demonstrate ares treatment means for mits [80%, 125%], if the n-inflamed lesion counts. |
|---|---|
| oximately om the mITT to the PP oo group are required ensure sufficient po ive treatment group are einflamed and non-ing each endpoint. Under equivalence and sup To allow erwise non-evaluable | in the mITT population |
| y with the protocol as | follows: |
| ta. ncomitant medication compliant w | Day $85 \pm 4$ days with no |
| | ese numbers, a sample vide approximately E/R ratio of least-square fined equivalence line veen inflamed and nor in inflammatory and eximately E/M ratio of least-square fined equivalence and nor in inflammatory and eximately E/M the mITT to the PP to group are required and ensure sufficient positive treatment group are inflamed and non-interest endpoint. Under the equivalence and supervise non-evaluable explacebo group). E/M with the protocol as the protocol window of ta. E/M with the protocol as the protocol window of ta. E/M comitant medication critical first protocol window of ta. E/M comitant medication critical first protocol window of ta. E/M comitant medication critical first protocol window of ta. |



# **Modified Intent-to-Treat Population (mITT)**

The mITT population will include all subjects in the PP population plus all randomized subjects who meet all inclusion/exclusion criteria, apply at least one dose of assigned product, and return for at least one post-Baseline evaluation.



# **Safety Population**

All subjects who are randomized and received IP will be included in the analysis of safety.

#### 7. STUDY EFFICACY VARIABLES

## **Primary Efficacy Endpoints**

The two co-primary efficacy endpoints are (1) the percent change from Baseline to Week 12 in the inflammatory (papules/pustules) lesion counts and (2) the percent change from Baseline to Week 12 in the non-inflammatory (open and closed comedones) lesion counts.

# **Secondary Efficacy Endpoint**

The secondary efficacy endpoint is the proportion of subjects who are considered a Clinical Success at Week 12, as defined by an IGA score that is at least 2 grades less than the Baseline assessment. That is, at Week 12, subjects with an IGA score of 4 at Baseline must achieve a score of 0, 1 or 2, subjects with an IGA score of 3 at Baseline must achieve a score of 0 or 1, and subjects with an IGA score of 2 at Baseline must achieve a score of 0 to be considered a Clinical Success.

A Clinical Failure is defined as an IGA score at Week 12 that is the same, higher or one grade lower than the Baseline IGA. Subjects who are discontinued due to lack of treatment effect or worsening condition will be considered Clinical Failures.

Tazarotene Cream 0.1%

Protocol /

0454-01-01/

## 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics, efficacy variables and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables with non-missing values, statistics will include number of observations, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS®, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

#### 8.1 Baseline Characteristics

# 8.1.1 Demographics Comparability of Treatment Groups

Baseline characteristics will be evaluated separately for the PP, mITT and Safety populations.

Demographic information collected at baseline includes the following:

- Age (years)
- Sex (Male/Female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- Baseline number of inflammatory lesions (i.e., papules and pustules)
- Baseline number of non-inflammatory lesions (i.e., open and closed comedones)
- Baseline number of nodulocystic lesions (i.e., nodules and cysts)
- Baseline IGA score

Summary tables by treatment group will be presented. Continuous variables will be summarized using descriptive statistics (number of observations, median, minimum, maximum, mean and standard deviation). Categorical variables will be summarized using frequencies and percentage. Baseline treatment comparisons will be presented using Chi-Square test for the categorical variables, and Analysis of Variance (ANOVA) for the continuous variables.

All data will be listed by treatment and patient.

Tazarotene Cream 0.1%

Protocol /

0454-01-01/

# 8.1.2 Medical History

At Visit 1 subjects will be questioned about personal medical history including acne history. The medical history will include a complete review of all current diseases and their respective durations and treatments.

Medical history data will be listed by treatment and patient.

## **8.1.3 Concomitant Medications**

At Visit 1, subjects will be questioned about current and prior concomitant medication use over the previous 6 months. At Visit 2, Visit 3 and Visit 4 subjects will be questioned about ongoing or new concomitant medication use

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and patient.

# 8.1.4 Pregnancy Test

All females of childbearing potential will have a urine pregnancy test performed at each Scheduled visit. All females of childbearing potential will have a urine pregnancy test performed at Visit 1 (Baseline), Visit 2, Visit 3, and Visit 4 (or early termination).

Pregnancy test results will be listed by treatment and patient.

## **8.2** Efficacy Analyses

# 8.2.1 Primary Efficacy Analysis

## **Therapeutic Bioequivalence Analysis**

The primary measure of therapeutic equivalence will be evaluated using the PP population, with results in the mITT population being supportive.

The following Statistical Analysis Method is recommended by OGD for equivalence testing for a continuous variable:

The compound hypothesis to be tested is:

$$H_0$$
:  $\mu T/\mu R < \theta 1$  or  $\mu T/\mu R > \theta 2$  versus

Tazarotene Cream 0.1%

Protocol /

0454-01-01/

$$H_A$$
:  $\theta 1 \le \mu T / \mu R \le \theta 2$ 

where  $\mu T$  = mean percent change from baseline of test treatment, and  $\mu R$  = mean percent change from baseline of reference treatment

Under the assumptions of normally distributed data, the adjusted 90% confidence interval will be calculated for the Test/Reference ratio of the mean percent change from Baseline in inflammatory and non-inflammatory lesion counts using an iterative procedure similar to Fieller's method. ANOVA with treatment and site as fixed effects in the model will be conducted on the mean percent change from Baseline to Week 12 in the inflammatory (papules/pustules) lesion counts and non-inflammatory (open and closed comedones) lesion counts. If the adjusted 90% confidence intervals for the least-squares mean Test/Reference ratios are within 80-125% for both co-primary endpoints, then therapeutic equivalence of the Test to Reference product will be considered to have been demonstrated.

To declare therapeutic equivalence of the Test product to the Reference product, therapeutic equivalence must be demonstrated for only the primary endpoints in the PP population.

# **Superiority to Placebo Analysis**

The primary measure of superiority will be evaluated using the mITT population, using LOCF for missing efficacy values. The results in the PP population will be considered supportive.

The superiority of the Test and Reference products over Placebo is concluded if these treatments' mean percent changes from Baseline in inflamed and non-inflamed lesion counts at Week 12 are statistically superior to that of the Placebo at the 5% significance level (p < 0.05, two-sided). The superiority of Test and Reference treatments over the Placebo will be evaluated in the same ANOVA model for Test vs. Placebo and Reference vs. Placebo.

To declare superiority of the Test and Reference products over Placebo, their superiority must be demonstrated for only the primary endpoint in the mITT population.

# 8.2.2 Secondary Efficacy Analyses

The PP population will be used for analysis of therapeutic equivalence and the mITT population will be used for analyses of superiority.

## Therapeutic Bioequivalence Analysis

Tazarotene Cream 0.1%

Protocol /

0454-01-01/

Based on the usual method used in OGD for binary outcomes, the 90% confidence interval for the difference in success proportions between test and reference treatment should be contained within [-0.20, +0.20] in order to establish equivalence.

The compound hypothesis to be tested is:

$$H_0: P_T - P_R < -.20 \text{ or } P_T - P_R > .20 \text{ versus}$$

$$H_A: -.20 \le P_T - P_R \le .20$$

where  $P_T$  = success rate of test treatment

 $P_R$  = success rate of reference treatment.

Let

 $n_T$  = sample size of test treatment group

 $cn_T$ = number of subjects considered as clinical success in test treatment group

 $n_R$  = sample size of reference treatment group

 $cn_R$  = number of subjects considered as clinical success in reference treatment group

$$\hat{P}_T = c n_T / n_T$$
  $\hat{P}_R = c n_R / n_R$ , and

$$se = (\widehat{P}_T (1 - \widehat{P}_T)/n_T + (\widehat{P}_R (1 - \widehat{P}_R)/n_R)^{1/2})$$

The 90% confidence interval for the difference in proportions between test and reference will be calculated as follows, using Yates' correction:

$$L = (\hat{P}_T - \hat{P}_R) - 1.645 se - (1/n_T + 1/n_R)/2$$

$$U = (\hat{P}_T - \hat{P}_R) + 1.645 se + (1/n_T + 1/n_R)/2$$

For the proportion of Clinical Success, if the 90% confidence interval (with Yates' Correction factor) of the difference between the proportion of subjects considered a Clinical Success in the Test and the Reference product groups at Week 12 is contained within -20% to +20%, then therapeutic equivalence of the Test to Reference product will be considered supported for the secondary endpoint.

# **Superiority to Placebo Analysis**

The analyses for superiority will be conducted using the mITT population and LOCF.

For the determination of superiority, the proportion of subjects considered a Clinical Success at Week 12 in the Test and Reference product groups will each be compared to the proportion of

4/26/2017

# Tazarotene Cream 0.1%

Protocol /

0454-01-01/

subjects considered as Clinical Success in the Placebo group.

If the proportion of subjects showing Clinical Success in the Test and Reference groups is statistically significantly greater (p < 0.05; using Cochran-Mantel-Haenszel exact test stratified by clinical site)) than the Clinical Success seen in the Placebo group then superiority will be concluded.

A summary table with frequency and percentage of the proportion of Clinical Success by treatment group will be presented.

# 8.2.3 Treatment-by-Site Interaction and Pooling of Clinical Sites

As this is a multiple-site study, the interaction of treatment-by-site may be evaluated in the ANOVA model for evaluations involving the primary efficacy endpoint.

If no treatment-by-site interaction is identified with the primary endpoint then no adjustment will be made to any efficacy analysis and treatment-by site interaction will not be included as a term in the statistical models for evaluating therapeutic equivalence and superiority.

## 8.3 Safety Analysis

All safety analyses will be based on the Safety Population.

## 8.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 18.1 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, relationship to the IP, action taken and outcome.

In each of the following categories, the total number and percentage of subjects with 1) at least one AE, 2) discontinued study drug due to AEs, 3) AE severity and AEs related to the IP, 4) serious AEs and death will be summarized separately by treatment groups.

A summary table of the number and percent of subjects with AEs by system organ class, preferred term, and treatment group will be presented. Each patient will be counted only once within each preferred term.

# Tazarotene Cream 0.1%

Protocol /

0454-01-01/

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment group will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to the IP, and treatment group will be presented. Relationship to a study drug will be classified as "Suspected" or "Not Suspected".

Should sufficient data exist, adverse event frequencies will be compared between treatments using Fisher's exact test.

# 8.3.2 Application Site Reactions

At Visits 1, 2, 3 and 4 the Investigator will evaluate the patient for local application site reactions based on the scale provided in Appendix B:

Signs and Symptoms recorded at each visit will be compared between treatment groups. Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) comparing the application site reactions for each treatment group will be presented by visit.

A frequency summary table comparing the application site reactions for each treatment group will be presented by visit.

## 8.3.3 Vital Signs

The patient's vital signs (pulse, blood pressure, temperature and respiration rate) will be recorded at Visit 1 and Visit 4.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit for non-missing values.

All data will be listed by treatment and patient.

## **8.4 Multiple Comparisons**

No multiple comparison adjustment will be made in this study.

## 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available

# Tazarotene Cream 0.1%

Protocol /

0454-01-01/

data. Subjects with missing data will be excluded only from analyses for which data are not available, including denominators.

Subjects discontinued early for reasons other than lack of treatment effect or worsening condition will be excluded from the PP population and included in the mITT population using Last Observation Carried Forward (LOCF), provided they administered at least one dose of randomized IP and completed at least one post-dose evaluation.

# 8.6 Interim Analyses

There is no interim analysis planned in this study.

# 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

| Fougera Pharmaceuticals Inc. | | |
|------------------------------|------------|-------------|
| Tazarotene Cream 0.1% | Protocol / | 0454-01-01/ |

# TABLE, LISTING AND FIGURE SHELLS

T16.1.9.1 Summary of Discontinued Subjects (Safety Population)

| Subjects | Test | Reference | Placebo | Total |
|--------------------------|------|-----------|---------|-------|
| Randomized | xxx | XXX | xxx | XXX |
| Completed Study | xxx | XXX | xxx | XXX |
| Terminated Early | xxx | XXX | xxx | XXX |
| Early Termination Reason | | | | |
| Administrative reasons | xxx | XXX | xxx | XXX |
| Lack of efficacy | xxx | XXX | xxx | xxx |
| Lost to Follow-Up | xxx | XXX | XXX | XXX |
| etc. | | | | |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

0454-01-01/

T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Test | Reference | Placebo | Total |
|-----------------------------------------|------|-----------|---------|-------|
| Total Subjects with Protocol Deviations | XXX | XXX | XXX | XXX |
| Total Deviations | XXX | XXX | XXX | XXX |
| Lost to follow up | XXX | XXX | XXX | XXX |
| Outside visit window | xxx | XXX | XXX | XXX |
| Missed Visit | xxx | XXX | xxx | XXX |
| Restricted Medication | xxx | XXX | XXX | XXX |
| etc | xxx | XXX | xxx | XXX |
| Other | xxx | XXX | XXX | XXX |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

T16.1.9.3.1 Summary of Subjects Excluded from Efficacy Analysis (Population Determination)

| | | Test | Reference | Placebo | Total |
|---|---|---|---|---|---|
| Randomized | Total | xxx | XXX | XXX | XXX |
| Safety Population | Total | xxx | XXX | xxx | xxx |
| Excluded from Safety | Did not received study product | XXX | xxx | xxx | XXX |
| | etc. | | | | |
| mITT Population | Total | xxx | XXX | xxx | xxx |
| Excluded from mITT | Did not received study product | XXX | xxx | xxx | XXX |
| | etc. | | | | |
| PP Population | Total | xxx | XXX | XXX | XXX |
| Excluded from Excluded from PP | Restricted Medication | XXX | XXX | xxx | xxx |
| | etc. | | | | |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ \SAS\OUT Created on: ddmmmyy hh:mm

| Protocol | / | . 0454-01-01/ |
|----------|---|---------------|

T16.1.9.3.2 Summary of Subjects Included in Analysis Population by Study Center

| | | | | PP | | | PP mITT | | | | Safety | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site<br>No. | Name | Total<br>Randomized | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

0454-01-01/

T16.1.9.4.1 Summary of Demographic Data (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Age (years) | n | xxx | xxx | XXX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | XX.X - XX.X | xx.x - xx.x | |
| Race | White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Black/African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Native Hawaiian or other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | American Indian or Alaska Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Sex | Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | X.XXXX |
| | Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | X.XXXX |
| | Not Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

N= number of subjects in the treatment group; n= number of subjects with data available; % is based on N

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 1 of 2

0454-01-01/

T16.1.9.4.2 Summary of Baseline Parameters (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Total Inflammatory Lesion Count | n | xxx | XXX | XXX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | XX.X - XX.X | xx.x - xx.x | xx.x - xx.x | |
| Total Non-Inflammatory Lesion Count | n | xxx | xxx | xxx | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Total Nodulocystic Lesion Count | n | XXX | XXX | XXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Investigator Global Assessment | Clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | X.XXXX |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

Note: N= number of subjects in the treatment group; n= number of subjects with data available; % is based on N

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 2 of 2

Similar tables will be created for T16.1.9.5.1, T16.1.9.5.2, T16.1.9.6.1 and T16.1.9.6.2

T16.1.9.5.1 Summary of Demographic Data (modified Intent-to-Treat Population)

T16.1.9.5.2 Summary of Baseline Parameters (modified Intent-to-Treat Population)

T16.1.9.6.1 Summary of Demographic Data (Per-Protocol Population)

T16.1.9.6.2 Summary of Baseline Parameters (Per-Protocol Population)

0454-01-01/

T16.1.9.7.1 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Inflammatory Lesion Count) (Per-Protocol Population)

| | | Test | Reference | Placebo | Overall |
|---|---|---|---|---|---|
| | Statistic | (N = xxx) | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ |
| Baseline | n | xxx | xxx | xxx | xxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | XX.X - XX.X | xx.x - xx.x | xx.x - xx.x |
| Week 12 | n | xxx | XXX | xxx | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | XX.X - XX.X | xx.x - xx.x | xx.x - xx.x |
| Percent Change from Baseline | n | XXX | XXX | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |

N= number of subjects in the treatment group; n= number of subjects with data available;

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC  $^{\! (\! )}$  (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

T16.1.9.7.2 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Inflammatory Lesion Count) (modified Intent-to-Treat Population)

| | | Test | Reference | Placebo | Overall |
|---|---|---|---|---|---|
| | Statistic | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ |
| Baseline | n | XXX | XXX | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Week 12 | n | XXX | XXX | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Percent Change from Baseline | n | XXX | XXX | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |

N= number of subjects in the treatment group; n= number of subjects with data available;

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

# T16.1.9.8.1 Summary of Analysis Results of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Inflammatory Lesion Count between Treatment Groups)

| <b>Equivalence: P</b> | er-Protocol Population | | | |
|---|---|---|---|---|
| | | | Difference Between Trea | tments |
| Treatment | Number of | | Test-to-Reference | ence |
| Group | Subjects (N) | LSMeans | Ratio | 90% CI Evaluation |
| Test | XXX | XXX.X | | |
| Reference | XXX | XXX.X | XX.X | xx.x - xx.x |

## **Superiority: modified Intent-to-Treat Population**

| | | | | Treatment vs. Placebo | | | |
|---|---|---|---|---|---|---|---|
| | | | | | Std Err | | |
| Treatment | Number of | | Std Err | LSMeans | LSMeans | | |
| Group | Subjects (N) | LSMeans | LSMeans | Difference | Difference | 95% CI | P-value |
| Placebo | xxx | XXX.X | XXX.X | | | | |
| Test | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |
| Reference | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |

The 90% confidence interval for the test-to-reference ratio was calculated using a procedure similar to Fieller's method.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

# T16.1.9.8.2 Summary of Supportive Analysis Results of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Inflammatory Lesion Count between Treatment Groups)

| | | | Difference Between Trea | tments |
|---|---|---|---|---|
| Freatment | Number of | | Test-to-Reference | |
| Group | Subjects (N) | LSMeans | Ratio | 90% CI Evaluation |
| Γest | XXX | XXX.X | | |
| Reference | XXX | XXX.X | XX.X | xx.x - xx.x |

## **Superiority: Per-Protocol Population**

| | | | | Treatment vs. Placebo | | | |
|---|---|---|---|---|---|---|---|
| | | | | | Std Err | | |
| Treatment | Number of | | Std Err | LSMeans | LSMeans | | |
| Group | Subjects (N) | LSMeans | LSMeans | Difference | Difference | 95% CI | P-value |
| Placebo | xxx | XXX.X | XXX.X | | | | |
| Test | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |
| Reference | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |

The 90% confidence interval for the test-to-reference ratio was calculated using a procedure similar to Fieller's method.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

T16.1.9.9.1 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Non-Inflammatory Lesion Count) (Per-Protocol Population)

| | | Test | Reference | Placebo | Overall |
|---|---|---|---|---|---|
| | Statistic | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ |
| Baseline | n | XXX | XXX | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Week 12 | n | xxx | xxx | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Range | XX.X - XX.X | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Percent Change from Baseline | n | xxx | XXX | XXX | XXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |

N= number of subjects in the treatment group; n= number of subjects with data available;

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

T16.1.9.9.2 Descriptive Summary of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Non-Inflammatory Lesion Count) (modified Intent-to-Treat Population)

| | | Test | Reference | Placebo | Overall |
|---|---|---|---|---|---|
| | Statistic | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ |
| Baseline | n | XXX | xxx | XXX | xxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | XX.X - XX.X | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| Week 12 | n | xxx | xxx | XXX | xxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | XX.X - XX.X | xx.x - xx.x | xx.x - xx.x |
| Percent Change from Baseline | n | xxx | XXX | XXX | xxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |

N= number of subjects in the treatment group; n= number of subjects with data available;

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

# T16.1.9.10.1 Summary of Analysis Results of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Non-Inflammatory Lesion Count between Treatment Groups)

| <b>Equivalence:</b> P | Equivalence: Per-Protocol Population | | | |
|---|---|---|---|---|
| | | Difference Between Treatments | | |
| Treatment | Number of | Test-to-Reference | | |
| Group | Subjects (N) | LSMeans | Ratio | 90% CI Evaluation |
| Test | XXX | XXX.X | | |
| Reference | XXX | XXX.X | XX.X | xx.x - xx.x |

## **Superiority: modified Intent-to-Treat Population**

| | | | | | Treatment vs. Placebo | | |
|---|---|---|---|---|---|---|---|
| | | | | | Std Err | | |
| Treatment | Number of | | Std Err | LSMeans | LSMeans | | |
| Group | Subjects (N) | LSMeans | LSMeans | Difference | Difference | 95% CI | P-value |
| Placebo | xxx | XXX.X | XXX.X | | | | |
| Test | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |
| Reference | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |

The 90% confidence interval for the test-to-reference ratio was calculated using a procedure similar to Fieller's method.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

# T16.1.9.10.2 Summary of Supportive Analysis Results of Co-Primary Efficacy Endpoint (Percent Change from Baseline in Non-Inflammatory Lesion Count between Treatment Groups)

| Treatment<br>Group | Number of<br>Subjects (N) | | eatments | |
|---|---|---|---|---|
| | | LSMeans | Ratio | 90% CI Evaluation |
| Test | XXX | XXX.X | | |
| Reference | XXX | XXX.X | XX.X | xx.x - xx.x |

## **Superiority: Per-Protocol Population**

| | | | | Treatment vs. Placebo | | | |
|---|---|---|---|---|---|---|---|
| | | | | | Std Err | | |
| Treatment | Number of | | Std Err | LSMeans | LSMeans | | |
| Group | Subjects (N) | LSMeans | LSMeans | Difference | Difference | 95% CI | P-value |
| Placebo | XXX | XXX.X | XXX.X | | | | |
| Test | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |
| Reference | xxx | XXX.X | XXX.X | XXX.X | XXX.X | xx.x - xx.x | X.XXXX |

The 90% confidence interval for the test-to-reference ratio was calculated using a procedure similar to Fieller's method.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm
0454-01-01/

# T16.1.9.11 Summary of Analysis Results of Secondary Efficacy Endpoint (Proportion of Clinical Successes Between Treatment Groups)

| Equivalence: Per-Protocol Population | | | | | |
|---|---|---|---|---|---|
| | | | | Difference B | Setween Treatments |
| Treatment | Number of | Number of<br>Treatment | Proportion of<br>Treatment | | |
| Group | Subjects (N) | Successes (n) | Successes (%) | Difference | 90% CI Evaluation |
| Test | XXX | xxx | xx.x% | | |
| Reference | xxx | xxx | XX.X% | xx.x% | xx.x - xx.x |

#### **Superiority: modified Intent-to-Treat Population**

| | | Number of | Proportion of | |
|-----------|--------------|---------------|---------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | xx.x% | |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm

0454-01-01/

**T16.1.9.12 Overall Summary of Adverse Events** (Safety Population)

| Description | Test<br>N (%) | Reference<br>N (%) | Placebo<br>N (%) | Total<br>N (%) |
|---|---|---|---|---|
| Subjects Randomized | xxx | xxx | xxx | xxx |
| Subjects with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued study drug due to above AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | XXX | XXX | XXX | XXX |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Suspected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suspected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

SAS\OUT Path: L:\Studies Sas Codes\Clinical Trial\

Created on: ddmmmyy hh:mm

## T16.1.9.13 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| | | Te<br>(N = | | | erence<br>= xxx) | | Placebo<br>N = xxx) | Fisher's |
|---|---|---|---|---|---|---|---|---|
| Body System | MedDRA Term | Events | Subjects | Events | Subjects | Events | Subjects | P-value |
| Patient with at least one AE | Total | Xx | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| Ear and labyrinth<br>disorders | Ear pain | Xx | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| | etc. | | | | | | | |

etc.

Comparison of treatment groups is with respect to the number of subjects with at least one occurrence of the AE.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

T16.1.9.14 Summary of Frequency for AEs Occurring in at Least 5% of Subjects by Body System (Safety Population)

0454-01-01/

T16.1.9.15 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| | | | Test # Events (N=xx) | | | Reference # Events (N=xx) | | | Placebo<br># Events<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Total AEs | Total AEs | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Hypoacusis | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

etc.

N = Total number of events in each treatment group; Percentage is based on total number of events.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

T16.1.9.16 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| | | Test # Events (N=xx) | | Reference # Events (N=xx) | | Placebo<br># Events<br>(N=xx) | |
|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Suspected | Not Suspected | Suspected | Not Suspected | Suspected | Not Suspected |
| Total AEs | Total AEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth | Ear pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| disorders | Hypoacusis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | etc. | | | | | | |

etc.

N = Total number of events in each treatment group; Percentage is based on total number of events.

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

## T16.1.9.17 Summary of Frequency of Serious Adverse Events (Safety Population)

| | | Test | Reference | Placebo |
|---|---|---|---|---|
| Body System | MedDRA Term | # Events | # Events | # Events |
| Injury, poisoning and procedural complications | Alcohol poisoning | XX | XX | XX |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

T16.1.9.18 Summary of Application Site Reaction (Safety Population)

| Signs and | | | Test | Reference | Placebo |
|---|---|---|---|---|---|
| Symptoms | Visit | Statistic | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | (N = xxx) |
| Erythema | 1 | n | xxx | XXX | xxx |
| | | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | | Median | XX.X | XX.X | XX.X |
| | | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| | 2 | | | | |
| | 3 | | | | |
| | 4/ET | | | | |

Dryness

Burning/Stinging

Erosion

Edema

Pain

Itching

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

## T16.1.9.19 Summary of Frequency of Application Site Reaction (Safety Population)

| Signs and | | | Test | Reference | Placebo |
|---|---|---|---|---|---|
| Symptoms | Visit | Statistic | (N = xxx) | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | (N = xxx) |
| Erythema | 1 | Absent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Mild | xxx (xx.x%) | xxx(xx.x%) | xxx (xx.x%) |
| | | Moderate | xxx (xx.x%) | xxx(xx.x%) | xxx (xx.x%) |
| | | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 2 | | | | |
| | 3 | | | | |
| | 4/ET | | | | |

Dryness

Burning/Stinging

Erosion

Edema

Pain

Itching

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/ Protocol /

## T16.1.9.20 Summary of Vital Signs (Safety Population)

| Vital Signs | Visit | Statistic | Test (N = xxx) | Reference $(N = xxx)$ | Placebo<br>(N = xxx) |
|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | 1 | n | XXX | XXX | XXX |
| | | $Mean \pm SD$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | | Median | XXX.X | XXX.X | XXX.X |
| | | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| | 4/ET | | | | |

Diastolic Blood Pressure (mmHg)

Pulse Rate (beats/min)

Respiration Rate (breaths/min)

Temperature (F)

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.1 Listing of Discontinued Subjects

| Treatment | Patient | Discontinuation | | _ |
|-----------|-----------|-------------------|------------|---|
| Group | Number | Reason | Population | |
| Test | xx - xxxx | Withdrew Consent | Safety | |
| | xx - xxxx | Lost to Follow-up | Safety | |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.2 Listing of Protocol Deviations

| Treatment | Patient | | |
|-----------|-----------|-----------------------------------|------------|
| Group | Number | <b>Protocol Deviation Summary</b> | Population |
| Test | xx - xxxx | Outside Visit Window | Safety |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

## L16.2.3.1 Subjects Excluded from the Per-Protocol Population Data Set

| Treatment | Patient | Exclusion |
|-----------|-----------|-------------------------------------|
| Group | Number | Reason |
| Test | xx - xxxx | Patient did not meet IE criterion. |
| | xx - xxxx | Patient took prohibited medications |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm

### L16.2.3.2 Subjects Excluded from the Modified Intent-to-Treat Data Set

| Treatment<br>Group | Patient<br>Number | Exclusion<br>Reason |
|---|---|---|
| Test | xx - xxxx | Patient did not have at least one post-randomization evaluation |
| | xx - xxxx | Patient did not have at least one post-randomization evaluation |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)
Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)
Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

SAS\OUT Path: L:\Studies Sas Codes\Clinical Trial\

Created on: ddmmmyy hh:mm Page 1 of N

## L16.2.4.1 Listing of Demographic Data

| Treatment | Patient | | | | |
|---|---|---|---|---|---|
| Group | Number | Age | Sex | Ethnicity | Race |
| Test | xx - xxxx | 30 | Female | Not Hispanic or Latino | Black or African American |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\SAS\OUT

Created on: ddmmmyy hh:mm

### L16.2.4.2 Listing of Medical History

| Treatment | Patient | | | | | |
|---|---|---|---|---|---|---|
| Group | Number | Category | Reported Term | <b>Onset Date</b> | <b>End Date</b> | Ongoing |
| Test | XX - XXXX | Gynecologic | Menopause | 2003 | 2003 | |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

## L16.2.4.3 Listing of Concomitant Medications

**Test: Tazarotene Cream 0.1%** 

| Patient | Medication/ | | | | | |
|---|---|---|---|---|---|---|
| Number | Therapy Name | Dosage | Frequency | Route | Date | Indication |
| xx - xxxx | LISINOPRIL | 20 MG | QD | PO | yyyy-mm-dd/ | HYPERTENSION |

Note to programmer: table will continue for reference and placebo group

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/ Protocol /

## L16.2.5.1 Listing of Visit Date Information

| Treatment | Patient | Inform Consent | Inform Consent | | | |
|---|---|---|---|---|---|---|
| Group | Number | Date | Visit 1 | Visit 2 | Visit 3 | <b>Early Termination</b> |
| Test | xx - xxxx | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd |

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.5.2 Listing of Drug Administration

| Treatment | Patient | Date of | Date of | Total Doses | Dosing |
|---|---|---|---|---|---|
| Group | Number | First Dose | Last Dose | Applied | Compliance (%) |
| Test | xx - xxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX.X |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

### L16.2.6.1 Listing of Lesion Count

| Treatment<br>Group | Patient<br>Number | Visit | Total<br>Inflammatory<br>Lesion Count | Total<br>Non-Inflammatory<br>Lesion Count | Total<br>Nodulocystic<br>Lesion Count | Percent Change<br>from Baseline in<br>Total Inflammatory<br>Lesion Count | Percent Change from Baseline in Total Non-Inflammatory Lesion Count |
|---|---|---|---|---|---|---|---|
| Test | xx - xxxx | 1 | XX | XX | xx | XX | 0.00 |
| | | 2 | xx | xx | xx | xx | X.XX |
| | | 3 | XX | XX | XX | XX | X.XX |
| | | 4/ET | xx | xx | xx | XX | X.XX |

etc

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

L16.2.6.2 Listing of Investigator Global Assessment

| Treatment<br>Group | Patient<br>Number | Visit | IGA | Change from<br>Baseline | Success/<br>Failure |
|---|---|---|---|---|---|
| Test | xx - xxxx | 1 | XX | 0 | |
| | | 2 | XX | XX | |
| | | 3 | XX | XX | |
| | | 4/ET | XX | XX | Success |
| | xx - xxxx | 1 | XX | 0 | |
| | | 2 | XX | XX | |
| | | 3 | XX | XX | |
| | | 4/ET | XX | XX | Failure |
| | etc | | | | |

Reference Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.7.1 Listing of Adverse Events by Treatment Group

**Test: Tazarotene Cream 0.1%** 

| Patient | • • | | Relationship<br>to Investigational | · | | | | |
|---|---|---|---|---|---|---|---|---|
| Number | AE Term | Area | Date | Severity | Drug | Outcome | Other Action Taken | SAE? |
| xx - xxxx | Nervous system disorders/ headache/<br>Headache | No | yyyy-mm-dd /<br>yyyy-mm-dd | Mild | Not Suspected | Recovered | Drug withdrawn/ None | No |

Note to programmer: table will continue for reference and placebo group

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm

## L16.2.7.2 Listing of Application Site Reactions

| Treatment<br>Group | Visit | Erythema | Dryness | Burning<br>/Stinging | Erosion | Edema | Pain | Itching |
|---|---|---|---|---|---|---|---|---|
| Test | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
| | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
| | 4/ET | 0 | 0 | 0 | 1 | 0 | 0 | 2 |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

## L16.2.8.1 Listing of Pregnancy Test Results

| Treatment | Patient | | | | Visit 4 or |
|---|---|---|---|---|---|
| Group | Number | Visit 1 | Visit 2 | Visit 3 | <b>Early Termination</b> |
| Test | xx - xxxx | Negative | Negative | Negative | Negative |

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

0454-01-01/

## L16.2.8.2 Listing of Vital Signs

| Treatment<br>Group | Patient<br>Number | Visit | Systolic BP (mmHg) | Diastolic BP<br>(mmHg) | Pulse Rate<br>(beats/min ) | Respiration Rate (breaths/min) | Temperature<br>(F) |
|---|---|---|---|---|---|---|---|
| Test | xx - xxxx | 1 | 120 | 70 | 84 | 18 | 98.6 |
| | | 4/ET | 140 | 80 | 74 | 18 | 97 |

xx - xxxx

Reference

Placebo

Test: Tazarotene Cream 0.1% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.1% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

SAS\OUT

Created on: ddmmmyy hh:mm

#### **Tazarotene Cream 0.1%**

Protocol /

0454-01-01/

## APPENDIX A: Investigator's Global Assessment for Acne Vulgaris

To be eligible for participation in the study a subject must have a Baseline IGA score of 2, 3 or 4.

| Grade | Description |
|---|---|
| 0 | Clear skin with no inflammatory or non-inflammatory lesions |
| 1 | Almost clear; rare non-inflammatory lesions with no more than one small inflammatory lesion |
| 2 | Mild severity; greater than Grade 1; some non-inflammatory lesions with no more than a few inflammatory lesions (papules/pustules only, no nodular lesions) |
| 3 | Moderate severity; greater than Grade 2; up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than one small nodular lesion |
| 4 | Severe; greater than Grade 3; up to many non-inflammatory lesions and may have some inflammatory lesions, but no more than a few nodular lesions |
| 5 | Greater than Grade 4 |

#### **Tazarotene Cream 0.1%**

Protocol /

0454-01-01/

## **APPENDIX B: Application Site Reactions**

The following application site reactions will be evaluated at each visit based on the scale provided below:

Signs and Symptoms:

Erythema

Dryness

Burning/Stinging

**Erosion** 

Edema

Pain

Itching

## **Grading Scale:**

| Severity | <u>Grade</u> |
|----------|--------------------------------|
| Absent | 0 |
| Mild | 1 (slight, barely perceptible) |
| Moderate | 2 (distinct presence) |
| Severe | 3 (marked, intense) |

| Tazarotene Cream 0.1% | Protocol / | 0454-01-01/ |
|-----------------------|------------|-------------|

| 1 azarotene Cream 0.1% Protocol/ 0454-01-01/ | Tazarotene Cream 0.1% | Protocol / | 0454-01-01/ |
|---|---|---|---|
|---|---|---|---|

